CLINICAL TRIAL: NCT00005515
Title: Mutations, Hormone Therapy (HRT) and Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5033; R01HL060739 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2005-07

CONDITIONS: Cardiovascular Diseases; Venous Thromboembolism; Postmenopause
MeSH Terms: conditions — Cardiovascular Diseases; Venous Thromboembolism

SUMMARY:
To assess the interaction between hormone replacement therapy and the prothrombotic mutations, Factor V Leiden and the recently described prothrombin mutation (20210A) on the incidence of venous thromboembolism (VTE) in a population-based case-control study conducted at Group Health Cooperative of Puget Sound (GHC).

DETAILED DESCRIPTION:
BACKGROUND:

Epidemiologic studies have identified Factor V Leiden as the most common cause of heritable thrombophilia, a prothrombotic mutation associated with a 5 to 7-fold increase in the risk of venous thromboembolism (VTE). In pre-menopausal women, the use of oral contraceptives is associated with a 4-fold increase in VTE risk, and the joint effects of oral contraceptive use and Factor V Leiden carriership increase the VTE risk of by a factor of 35. Recently, the results of several observational studies and randomized clinical trials suggest that in post-menopausal women, the use of hormone replacement therapy is associated with a 3-fold increase in VTE risk. Whether post-menopausal women with prothrombotic mutations experience a similar 20-fold increase in risk when they take post-menopausal hormones remains unknown.

DESIGN NARRATIVE:

In this case-control study, post-menopausal women with a first episode of objectively confirmed venous thromboembolism, and population-based controls were identified and recruited from the GHC enrollment files. Controls were frequency matched to the cases on age and calendar-year. Data collection included a review of ambulatory medical record and a telephone interview. The GHC computerized pharmacy database was used to assess exposure to hormone replacement therapy. A venous blood specimen was obtained from consenting subjects, processed into aliquots of white cells, plasma, and red cells, and stored at 70 degrees C prior to laboratory analysis. DNA was extracted from white cells, and molecular genotyping assays were conducted to assess carriership of prothrombotic mutations.

ELIGIBILITY:
No eligibility criteria

Ages: 30 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Psaty — University of Washington

REFERENCES:
- [Background] Psaty BM, Smith NL, Lemaitre RN, Vos HL, Heckbert SR, LaCroix AZ, Rosendaal FR. Hormone replacement therapy, prothrombotic mutations, and the risk of incident nonfatal myocardial infarction in postmenopausal women. JAMA. 2001 Feb 21;285(7):906-13. doi: 10.1001/jama.285.7.906. PMID 11180734
- [Background] Klungel OH, Heckbert SR, Longstreth WT Jr, Furberg CD, Kaplan RC, Smith NL, Lemaitre RN, Leufkens HG, de Boer A, Psaty BM. Antihypertensive drug therapies and the risk of ischemic stroke. Arch Intern Med. 2001 Jan 8;161(1):37-43. doi: 10.1001/archinte.161.1.37. PMID 11146696
- [Background] Psaty BM, Furberg CD, Pahor M, Alderman M, Kuller LH. National guidelines, clinical trials, and quality of evidence. Arch Intern Med. 2000 Sep 25;160(17):2577-80. doi: 10.1001/archinte.160.17.2577. No abstract available. PMID 10999970
- [Background] Psaty BM, Smith NL, Heckbert SR, Vos HL, Lemaitre RN, Reiner AP, Siscovick DS, Bis J, Lumley T, Longstreth WT Jr, Rosendaal FR. Diuretic therapy, the alpha-adducin gene variant, and the risk of myocardial infarction or stroke in persons with treated hypertension. JAMA. 2002 Apr 3;287(13):1680-9. doi: 10.1001/jama.287.13.1680. PMID 11926892
- [Background] Psaty BM, Doggen C, Vos HL, Vandenbroucke JP, Rosendaal FR. Association of the alpha-adducin polymorphism with blood pressure and risk of myocardial infarction. J Hum Hypertens. 2000 Feb;14(2):95-7. doi: 10.1038/sj.jhh.1000943. PMID 10723114
- [Background] Psaty BM, Rennie D. Stopping medical research to save money: a broken pact with researchers and patients. JAMA. 2003 Apr 23-30;289(16):2128-31. doi: 10.1001/jama.289.16.2128. No abstract available. PMID 12709471
- [Background] Reiner AP, Heckbert SR, Vos HL, Ariens RA, Lemaitre RN, Smith NL, Lumley T, Rea TD, Hindorff LA, Schellenbaum GD, Rosendaal FR, Siscovick DS, Psaty BM. Genetic variants of coagulation factor XIII, postmenopausal estrogen therapy, and risk of nonfatal myocardial infarction. Blood. 2003 Jul 1;102(1):25-30. doi: 10.1182/blood-2002-07-2308. Epub 2002 Nov 27. PMID 12456499
- [Background] Bis JC, Smith NL, Psaty BM, Heckbert SR, Edwards KL, Lemaitre RN, Lumley T, Rosendaal FR. Angiotensinogen Met235Thr polymorphism, angiotensin-converting enzyme inhibitor therapy, and the risk of nonfatal stroke or myocardial infarction in hypertensive patients. Am J Hypertens. 2003 Dec;16(12):1011-7. doi: 10.1016/j.amjhyper.2003.07.018. PMID 14643574
- [Background] Doggen CJ, Lemaitre RN, Smith NL, Heckbert SR, Psaty BM. HMG CoA reductase inhibitors and the risk of venous thrombosis among postmenopausal women. J Thromb Haemost. 2004 May;2(5):700-1. doi: 10.1111/j.1538-7836.2004.00696.x. No abstract available. PMID 15099273
- [Background] Smith NL, Heckbert SR, Lemaitre RN, Reiner AP, Lumley T, Weiss NS, Larson EB, Rosendaal FR, Psaty BM. Esterified estrogens and conjugated equine estrogens and the risk of venous thrombosis. JAMA. 2004 Oct 6;292(13):1581-7. doi: 10.1001/jama.292.13.1581. PMID 15467060
- [Background] Tirschwell DL, Smith NL, Heckbert SR, Lemaitre RN, Longstreth WT Jr, Psaty BM. Association of cholesterol with stroke risk varies in stroke subtypes and patient subgroups. Neurology. 2004 Nov 23;63(10):1868-75. doi: 10.1212/01.wnl.0000144282.42222.da. PMID 15557504